CLINICAL TRIAL: NCT01735578
Title: Splanchnic Tissue Oxygenation During Enteral Feedings in Anemic Premature Infants at Risk for Necrotizing Enterocolitis
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 58673
Record Dates: First submitted 2012-11-22; First posted 2012-11-28 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2014-12

CONDITIONS: Anemia of Prematurity; Necrotizing Enterocolitis
Keywords: splanchnic oxygen saturations
MeSH Terms: conditions — Anemia; Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Premature infants with anemia: Inpatient premature infants at the University of Utah Neonatal Intensive Care Unit (NICU) with Hct < or = to 28 who are being fed and are stable.

SUMMARY:
Necrotizing enterocolitis (NEC) is the most common gastrointestinal emergency encountered in the newborn intensive care unit and represents a significant cause of morbidity and mortality in infants born prematurely. Among possible risk factors, a strong association between elective RBC transfusions in premature infants with anemia and the subsequent development of NEC has been consistently observed (6-11). However, a significant (and increasing) number of VLBW infants with anemia are managed with erythropoiesis stimulating agents (such as Epo) and iron and do not receive RBC transfusions during their hospital stay. The present study proposes to study this particular group of VLBW infants that remain with low (<28 %) hematocrit while receiving full enteral feedings.

The investigators hypothesize that significant anemia in VLBW infants will be associated with a baseline low cerebro-splanchnic oxygenation ratio (CSOR) (<0.75) as measured by NIRS, and that nasogastric feedings (NGF) in those particular patients will lead to further decreased splanchnic oxygenation. The investigators further postulate that CSOR values will be significantly lower among VLBW that develop NEC as compared to infants that do not.

DETAILED DESCRIPTION:
Necrotizing enterocolitis (NEC) is the most common gastrointestinal emergency encountered in the newborn intensive care unit and represents a significant cause of morbidity and mortality in infants born prematurely. This disease complicates the management of approximately 6 - 10% of very low birthweight (VLBW) infants and can result in significant feeding intolerance, intestinal perforation and/or death despite aggressive treatment (1). The sequence of events leading to NEC appears to be multifactorial and complex (2,3). While epidemiologic studies have identified multiple factors that appear to increase an infant's risk for the development of NEC, other than prematurity, no single predictive risk factor has been clearly delineated (4,5).

Among possible risk factors, a strong association between elective RBC transfusions in premature infants with anemia and the subsequent development of NEC has been consistently observed (6-11). Possible explanations for transfusion-associated NEC have been proposed: 1) the physiological impact of anemia that can initiate a cascade of events leading to ischemic-hypoxemic mucosal gut injury predisposing to NEC (10); 2) increased splanchnic blood flow following RBC transfusion leading to reperfusion injury of gut mucosa.

A significant (and increasing) number of VLBW infants with anemia are managed with erythropoiesis stimulating agents (such as Epo) and iron and do not receive RBC transfusions during their hospital stay. The present study proposes to study this particular group of VLBW infants that remain with low (<28 %) hematocrit while receiving full enteral feedings.

Near Infrared Spectroscopy (NIRS) is a non-invasive, FDA approved, bedside technology that allows determination of regional oxygen saturations (rSO2) in tissues such as the gut mesentery. Using NIRS, the oxygenation status of hemoglobin in tissues located 2-4 cm below the skin can be determined and recorded continuously (12). For instance, Dave et al. used NIRS to demonstrate that splanchnic rSO2, but not cerebral rSO2, increases after feeds in the stable prematurely born infant tolerating full bolus orogastric feedings (13). Of importance, the average hematocrit in this study group was 37% (±7) and therefore these babies had no significant anemia.

While no normative values exist for mesenteric rSO2 in premature infants, recent studies have explored NIRS use in determining gut hypoxia and ischemia (14). Abdominal NIRS was used to detect alterations of intestinal rSO2 and perfusion in premature piglets that developed NEC (15). In a prospective cohort study of 40 neonates with medical or surgical acute intraabdominal pathology, a cerebro-splanchnic oxygenation ratio (CSOR) of less than 0.75 predicted gut ischemia with 90% sensitivity (16).

While these studies support a role for NIRS monitoring of mesenteric rSO2, it is not clear whether 1) VLBW with significant anemia have perturbations in intestinal oxygenation and perfusion, and 2) alterations in mesenteric rSO2 predict the development of NEC in VLBW infants.

We hypothesize that significant anemia in VLBW infants will be associated with a baseline low CSOR (<0.75) as measured by NIRS, and that nasogastric feedings (NGF) in those particular patients will lead to further decreased splanchnic oxygenation. We further postulate that CSOR values will be significantly lower among VLBW that develop NEC as compared to infants that do not.

ELIGIBILITY:
Inclusion Criteria:

1. Premature infants of ≤ 32 weeks gestational age
2. anemia (hematocrit of ≤ 28 %)
3. full enteral feedings
4. stable clinical condition (no mechanical ventilation, no vasopressors, no sepsis)
5. Age ≤ 12 weeks of life

Exclusion Criteria:

1. Lack of parental consent
2. Multiple congenital anomalies
3. unstable clinical condition (mechanical ventilation, vasopressors, sepsis)
4. Previous medical or surgical NEC (defined as ≥ Bell's Stage II disease)

Max Age: 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants admitted to the University of Utah NICU with significant anemia.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2012-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
cerebro-splanchnic oxygenation ratio (CSOR) measurements | 24 hours
  Stable premature infants who are being fed but have hematocrits lower than or equal to 28 will be continuously monitored using near-infrared spectroscopy (NIRS) in the cerebral and mesenteric regions for 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Baserga, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Yost CC. Neonatal necrotizing enterocolitis: diagnosis, management, and pathogenesis. J Infus Nurs. 2005 Mar-Apr;28(2):130-4. doi: 10.1097/00129804-200503000-00007. PMID 15785334
- [Background] Frost BL, Jilling T, Caplan MS. The importance of pro-inflammatory signaling in neonatal necrotizing enterocolitis. Semin Perinatol. 2008 Apr;32(2):100-6. doi: 10.1053/j.semperi.2008.01.001. PMID 18346533
- [Background] Neu J, Mshvildadze M, Mai V. A roadmap for understanding and preventing necrotizing enterocolitis. Curr Gastroenterol Rep. 2008 Oct;10(5):450-7. doi: 10.1007/s11894-008-0084-x. PMID 18799119
- [Background] Lemons JA, Bauer CR, Oh W, Korones SB, Papile LA, Stoll BJ, Verter J, Temprosa M, Wright LL, Ehrenkranz RA, Fanaroff AA, Stark A, Carlo W, Tyson JE, Donovan EF, Shankaran S, Stevenson DK. Very low birth weight outcomes of the National Institute of Child health and human development neonatal research network, January 1995 through December 1996. NICHD Neonatal Research Network. Pediatrics. 2001 Jan;107(1):E1. doi: 10.1542/peds.107.1.e1. PMID 11134465
- [Background] Hunter CJ, Upperman JS, Ford HR, Camerini V. Understanding the susceptibility of the premature infant to necrotizing enterocolitis (NEC). Pediatr Res. 2008 Feb;63(2):117-23. doi: 10.1203/PDR.0b013e31815ed64c. PMID 18091350
- [Background] Christensen RD, Lambert DK, Henry E, Wiedmeier SE, Snow GL, Baer VL, Gerday E, Ilstrup S, Pysher TJ. Is "transfusion-associated necrotizing enterocolitis" an authentic pathogenic entity? Transfusion. 2010 May;50(5):1106-12. doi: 10.1111/j.1537-2995.2009.02542.x. Epub 2009 Dec 29. PMID 20051059
- [Background] Mally P, Golombek SG, Mishra R, Nigam S, Mohandas K, Depalhma H, LaGamma EF. Association of necrotizing enterocolitis with elective packed red blood cell transfusions in stable, growing, premature neonates. Am J Perinatol. 2006 Nov;23(8):451-8. doi: 10.1055/s-2006-951300. Epub 2006 Sep 28. PMID 17009195
- [Background] Josephson CD, Wesolowski A, Bao G, Sola-Visner MC, Dudell G, Castillejo MI, Shaz BH, Easley KA, Hillyer CD, Maheshwari A. Do red cell transfusions increase the risk of necrotizing enterocolitis in premature infants? J Pediatr. 2010 Dec;157(6):972-978.e1-3. doi: 10.1016/j.jpeds.2010.05.054. Epub 2010 Jul 21. PMID 20650470
- [Background] Blau J, Calo JM, Dozor D, Sutton M, Alpan G, La Gamma EF. Transfusion-related acute gut injury: necrotizing enterocolitis in very low birth weight neonates after packed red blood cell transfusion. J Pediatr. 2011 Mar;158(3):403-9. doi: 10.1016/j.jpeds.2010.09.015. Epub 2010 Nov 10. PMID 21067771
- [Background] Singh R, Visintainer PF, Frantz ID 3rd, Shah BL, Meyer KM, Favila SA, Thomas MS, Kent DM. Association of necrotizing enterocolitis with anemia and packed red blood cell transfusions in preterm infants. J Perinatol. 2011 Mar;31(3):176-82. doi: 10.1038/jp.2010.145. Epub 2011 Jan 27. PMID 21273983
- [Background] El-Dib M, Narang S, Lee E, Massaro AN, Aly H. Red blood cell transfusion, feeding and necrotizing enterocolitis in preterm infants. J Perinatol. 2011 Mar;31(3):183-7. doi: 10.1038/jp.2010.157. Epub 2011 Jan 20. PMID 21252964
- [Background] Baserga MC, Gregory GA, Sola A. Cerebrovascular response in small preterm infants during routine nursery gavage feedings. Biol Neonate. 2003;83(1):12-8. doi: 10.1159/000067011. PMID 12566677
- [Background] Dave V, Brion LP, Campbell DE, Scheiner M, Raab C, Nafday SM. Splanchnic tissue oxygenation, but not brain tissue oxygenation, increases after feeds in stable preterm neonates tolerating full bolus orogastric feeding. J Perinatol. 2009 Mar;29(3):213-8. doi: 10.1038/jp.2008.189. Epub 2008 Nov 20. PMID 19020529
- [Background] Dani C, Pratesi S, Fontanelli G, Barp J, Bertini G. Blood transfusions increase cerebral, splanchnic, and renal oxygenation in anemic preterm infants. Transfusion. 2010 Jun;50(6):1220-6. doi: 10.1111/j.1537-2995.2009.02575.x. Epub 2010 Jan 22. PMID 20113454
- [Background] Gay AN, Lazar DA, Stoll B, Naik-Mathuria B, Mushin OP, Rodriguez MA, Burrin DG, Olutoye OO. Near-infrared spectroscopy measurement of abdominal tissue oxygenation is a useful indicator of intestinal blood flow and necrotizing enterocolitis in premature piglets. J Pediatr Surg. 2011 Jun;46(6):1034-40. doi: 10.1016/j.jpedsurg.2011.03.025. PMID 21683194
- [Background] Fortune PM, Wagstaff M, Petros AJ. Cerebro-splanchnic oxygenation ratio (CSOR) using near infrared spectroscopy may be able to predict splanchnic ischaemia in neonates. Intensive Care Med. 2001 Aug;27(8):1401-7. doi: 10.1007/s001340100994. PMID 11511955